CLINICAL TRIAL: NCT04572269
Title: Metabolomics of Obstructive Sleep Apnea
Acronym: MOSA
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: University of Iceland (Other)
Responsible Party: Sponsor
Other Study IDs: 835027
Record Dates: First submitted 2020-09-25; First posted 2020-10-01 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: Metabolomics; Biomarker; PAP; OSA Subtype; Personalized medicine
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, Plasma, Platelet Poor Plasma (PPP), Peripheral Blood Monocyte Cell (PBMC) and anticoagulated whole blood,
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with OSA: Female and male subjects with Obstructive Sleep Apnea (OSA) (AHI >5)
  Interventions: Other: No Intervention

INTERVENTIONS:
Other: No Intervention — This protocol does not involve an intervention of drug/device, diet, exercise or PAP compliance.

SUMMARY:
This is an R01 funded project that focuses on the utility of metabolomics as a biomarker for OSA. Aims 1 and 3 leverages banked samples previously collected from subjects with and without OSA at the University of Pennsylvania and University of Iceland. Aim 2 is a prospective study that will collect serum samples from OSA subjects at the University of Pennsylvania and the University of Iceland.

DETAILED DESCRIPTION:
The primary objective of Aim 2 is to conduct a prospective observational study to evaluate the metabolomic changes in response to six months of positive airway pressure (PAP) treatment among OSA patients. Newly diagnosed OSA patients (AHI>5) will undergo additional measurements including: accelerometer x one week (to inform the metabolomics), Type 2 home sleep test (to assist with OSA subtyping), next morning blood draw, 24-hour diet recall (to inform the metabolomics), questionnaires and PVT.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Male or female, aged 30-75 years old
4. In good general health as evidenced by medical history and diagnosed with Obstructive Sleep Apnea (defined as AHI>5)
5. Ability to use accelerometer, perform Type 2 sleep test at home and agree to use PAP treatment.
6. For females of reproductive potential: use of highly effective contraception for at least 1 month prior to screening and agreement to use such a method during study participation.

Exclusion Criteria:

1. Current use of PAP treatment or mandibular advancement device or INSPIRE device
2. Presence of active cancer treatment or heart failure (ejection fraction <40%)
3. Pregnancy or lactation
4. Known allergic reactions to components of the plastic (used in PAP mask)
5. Febrile illness within 2 weeks of signing consent
6. Current drug or alcohol abuse
7. Known diagnosis and treatment of diabetes because this will independently alter metabolomic results.
8. Previously drawn laboratory Hemoglobin A1C above normal range (indicative of diabetes).

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Prospective recruitment of female and male OSA subjects n=500/site: Site #1 is University of Pennsylvania; Site #2 is University of Iceland for a total of n=1000 cases.
Sampling Method: Probability Sample
Enrollment: 388 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2025-09-12 (Actual); Study Completion 2025-09-12 (Actual)

PRIMARY OUTCOMES:
Assess the utility of metabolomics to diagnose OSA and access whether these metabolomic signatures change with PAP treatment. | We anticipate prospective recruitment to be completed within 3.5 years with final analyses completed by year 4.
  New OSA patients, AHI>5 will be recruited. Since this is a real-world trial, compliance of PAP usage will vary from 0 to 100%. Thus, we will be able to assess not only what metabolomic changes occur with PAP usage but also whether there is a correlation to the amount of PAP usage. Metabolomics can be used as a biomarker that correlates with duration and frequency of PAP usage. This will then be correlated to subjective and objective measures of daytime sleepiness (questionnaires + PVT) and sleep fragmentation.

SECONDARY OUTCOMES:
Determine a metabolic signature that correlates with duration and frequency of PAP usage. This will then be correlated to subjective and objective measures of daytime sleepiness and sleep fragmentation. | We anticipate prospective recruitment to be completed within 3.5 years with final analyses completed by year 4.
  We will assess whether there is a specific metabolic signature that strongly associates with PAP adherence, potentially independent of the metabolites in Outcome 1. Identifying the set of metabolites with the strongest association with PAP usage will allow us to define an objective biomarker for quantifying PAP adherence. Moreover, the pathways implicated by these biomarkers are likely to allude to certain mechanisms of response.

OTHER OUTCOMES:
Evaluate whether the metabolomic response to PAP treatment is modified by degree of obesity. | We anticipate prospective recruitment to be completed within 3.5 years with final analyses completed by year 4.
  We will utilize conditional MSMs that estimate whether the effect of PAP varies with BMI.
Examine whether OSA symptom subtypes have a different metabolomic responses to PAP treatment. | We anticipate prospective recruitment to be completed within 3.5 years with final analyses completed by year 4.
  We will utilize conditional MSMs that estimate whether the effect of PAP varies across symptom subtypes.

CONTACTS AND LOCATIONS:
Overall Officials: Allan Pack, MBChB, PhD, Principal Investigator — University of Pennsylvania; Aalim Weljie, PhD, Principal Investigator — University of Pennsylvania
Locations (2):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States
- University of Iceland, Reykjavik, Iceland

IPD SHARING:
Plan to Share IPD: Yes
Study participant research data, which is for purposes of statistical analysis and scientific reporting, will be transmitted to and stored in REDcap. This will not include the participant's contact or identifying information. Rather, individual participants and their research data will be identified by a unique study identification number. The study data entry and study management systems used by clinical sites and by the University of Pennsylvania research staff will be secured and password protected. At the end of the study, all study databases will be de-identified and archived at figshare <https://figshare.com>.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will be available to research teams within 1 year following study completion.
Access Criteria: Data collected for this study will be analyzed and stored in figshare <https://figshare.com>. After the study is completed, the de-identified, archived data will be transmitted to and stored in figshare <https://figshare.com>, for use by other researchers including those outside of the study.
URL: http://figshare.com

REFERENCES:
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Lim DC, Pack AI. Obstructive Sleep Apnea: Update and Future. Annu Rev Med. 2017 Jan 14;68:99-112. doi: 10.1146/annurev-med-042915-102623. Epub 2016 Oct 5. PMID 27732789
- [Background] Duran-Cantolla J, Aizpuru F, Martinez-Null C, Barbe-Illa F. Obstructive sleep apnea/hypopnea and systemic hypertension. Sleep Med Rev. 2009 Oct;13(5):323-31. doi: 10.1016/j.smrv.2008.11.001. Epub 2009 Jun 9. PMID 19515590
- [Background] Mehra R, Benjamin EJ, Shahar E, Gottlieb DJ, Nawabit R, Kirchner HL, Sahadevan J, Redline S; Sleep Heart Health Study. Association of nocturnal arrhythmias with sleep-disordered breathing: The Sleep Heart Health Study. Am J Respir Crit Care Med. 2006 Apr 15;173(8):910-6. doi: 10.1164/rccm.200509-1442OC. Epub 2006 Jan 19. PMID 16424443
- [Background] Li M, Hou WS, Zhang XW, Tang ZY. Obstructive sleep apnea and risk of stroke: a meta-analysis of prospective studies. Int J Cardiol. 2014 Mar 15;172(2):466-9. doi: 10.1016/j.ijcard.2013.12.230. Epub 2014 Jan 10. No abstract available. PMID 24452224
- [Background] Yaggi HK, Concato J, Kernan WN, Lichtman JH, Brass LM, Mohsenin V. Obstructive sleep apnea as a risk factor for stroke and death. N Engl J Med. 2005 Nov 10;353(19):2034-41. doi: 10.1056/NEJMoa043104. PMID 16282178
- [Background] Gozal D, Jortani S, Snow AB, Kheirandish-Gozal L, Bhattacharjee R, Kim J, Capdevila OS. Two-dimensional differential in-gel electrophoresis proteomic approaches reveal urine candidate biomarkers in pediatric obstructive sleep apnea. Am J Respir Crit Care Med. 2009 Dec 15;180(12):1253-61. doi: 10.1164/rccm.200905-0765OC. Epub 2009 Sep 24. PMID 19797158
- [Background] Young T, Palta M, Dempsey J, Skatrud J, Weber S, Badr S. The occurrence of sleep-disordered breathing among middle-aged adults. N Engl J Med. 1993 Apr 29;328(17):1230-5. doi: 10.1056/NEJM199304293281704. PMID 8464434
- [Background] Schaffer JE. Lipotoxicity: when tissues overeat. Curr Opin Lipidol. 2003 Jun;14(3):281-7. doi: 10.1097/00041433-200306000-00008. PMID 12840659
- [Background] Taylor WM, Halperin ML. Effect of valine on the control of fatty acid synthesis in white adipose tissue of the rat. Can J Biochem. 1975 Oct;53(10):1054-60. doi: 10.1139/o75-145. PMID 1203753
- [Background] Gehrman P, Sengupta A, Harders E, Ubeydullah E, Pack AI, Weljie A. Altered diurnal states in insomnia reflect peripheral hyperarousal and metabolic desynchrony: a preliminary study. Sleep. 2018 May 1;41(5):zsy043. doi: 10.1093/sleep/zsy043. PMID 29522222
- [Background] Weljie AM, Newton J, Mercier P, Carlson E, Slupsky CM. Targeted profiling: quantitative analysis of 1H NMR metabolomics data. Anal Chem. 2006 Jul 1;78(13):4430-42. doi: 10.1021/ac060209g. PMID 16808451
- [Background] Sengupta A, Krishnaiah SY, Rhoades S, Growe J, Slaff B, Venkataraman A, Olarerin-George AO, Van Dang C, Hogenesch JB, Weljie AM. Deciphering the Duality of Clock and Growth Metabolism in a Cell Autonomous System Using NMR Profiling of the Secretome. Metabolites. 2016 Jul 27;6(3):23. doi: 10.3390/metabo6030023. PMID 27472375